CLINICAL TRIAL: NCT05069896
Title: A Bioequivalence Study of Injections of Mirikizumab Solution Using Investigational 1-mL and 2-mL Pre-Filled Syringes and Investigational 1-mL and 2-mL Autoinjectors in Healthy Participants
Brief Title: A Study to Compare Two Formulations of Mirikizumab (LY3074828) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 18139; I6T-MC-AMBX (Other: Eli Lilly and Company)
Record Dates: First submitted 2021-10-01; First posted 2021-10-06 (Actual); Results first posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02-04

CONDITIONS: Healthy
MeSH Terms: interventions — mirikizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mirikizumab - Prefilled Syringe (Experimental): Participants received 3 milliliter (mL) mirikizumab as 2 subcutaneous (SC) injections of 1 mL and 2 mL delivered via a prefilled syringe (PFS) to abdomen or arms or thighs.
  Interventions: Drug: Mirikizumab Prefilled Syringe
- Mirikizumab - Autoinjector (Experimental): Participants received 3 mL mirikizumab as 2 SC injections of 1 mL and 2 mL delivered an autoinjector (AI) to abdomen or arms or thighs.
  Interventions: Drug: Mirikizumab Autoinjector

INTERVENTIONS:
Drug: Mirikizumab Prefilled Syringe — Administered SC by prefilled syringe
  Other Names: LY3074828
  Arms: Mirikizumab - Prefilled Syringe
Drug: Mirikizumab Autoinjector — Administered SC by autoinjector
  Other Names: LY3074828
  Arms: Mirikizumab - Autoinjector

SUMMARY:
The main purpose of this study is to compare the amount of mirikizumab that gets into the blood stream and how long it takes the body to get rid of it, when given as a solution formulation via manual prefilled syringe or autoinjector. The information about any adverse effects experienced will be collected and the tolerability of mirikizumab will also be evaluated.

Screening is required within 28 days prior to the enrolment. For each participant, the total duration of the clinical trial will be about 17 weeks including screening.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males or non-pregnant females of childbearing or non-childbearing potential
* Have body mass index (BMI) within the range 18.0 to 32.0 kg/m2 (inclusive)

Exclusion Criteria:

* Must not show evidence of active or latent tuberculosis (TB)
* Must not have received live vaccine(s) (including attenuated live vaccines and those administered intranasally) within 8 weeks of screening, or intend to during the study
* Must not have been treated with steroids within 1 month of screening, or intend to during the study
* Must not have had a serious infection, or have been hospitalized or have received IV antibiotics for an infection within 12 weeks prior to Day 1
* Must not be immunocompromised
* Must not have received treatment with biologic agents (e.g. monoclonal antibodies, including marketed drugs) within 3 months or 5 half-lives (whichever is longer) prior to Day 1
* Must not have clinically significant multiple or severe drug allergies, or intolerance to topical corticosteroids, or severe post treatment hypersensitivity reactions
* Must not have had lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years
* Must not have had breast cancer within the past 10 years
* Must not have significant allergies to humanized monoclonal antibodies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - LabCorp CRU, Inc., Daytona Beach, Florida
  - QPS, Springfield, Missouri
  - Covance Dallas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang X, Otani Y, Payne CD, Morris NJ, Chua L, Escobar R, Wang S, Shi G. Pharmacokinetic Bridging Between an Autoinjector and a Prefilled Syringe Following Subcutaneous Administration of Mirikizumab in Healthy Participants. Adv Ther. 2025 Nov;42(11):5529-5546. doi: 10.1007/s12325-025-03335-z. Epub 2025 Sep 3. PMID 40900263

RESULTS

PARTICIPANT FLOW:
Groups:
- Mirikizumab Pre-filled Syringe (PFS) - Abdomen: Participants received 3 milliliter (mL) mirikizumab as 2 subcutaneous (SC) injections of 1 mL and 2 mL delivered via PFS in the abdomen.
- Mirikizumab PFS - Arm: Participants received 3 mL mirikizumab as 2 SC injections of 1 mL and 2 mL delivered via PFS to arms.
- Mirikizumab PFS - Thigh: Participants received 3 mL mirikizumab as 2 SC injections of 1 mL and 2 mL delivered via PFS to thighs.
- Mirikizumab Autoinjector (AI) - Abdomen: Participants received 3 mL mirikizumab as 2 SC injections of 1 mL and 2 mL delivered via AI to the abdomen.
- Mirikizumab AI - Arm: Participants received 3 mL mirikizumab as 2 SC injections of 1 mL and 2 mL delivered via AI to arms.
- Mirikizumab AI - Thigh: Participants received 3 mL mirikizumab as 2 SC injections of 1 mL and 2 mL delivered via AI to thighs.
Period: Overall Study
Arm/Group | Mirikizumab Pre-filled Syringe (PFS) - Abdomen | Mirikizumab PFS - Arm | Mirikizumab PFS - Thigh | Mirikizumab Autoinjector (AI) - Abdomen | Mirikizumab AI - Arm | Mirikizumab AI - Thigh
Started | 39 | 39 | 39 | 40 | 40 | 40
Received At Least One Dose of Study Drug | 39 | 39 | 39 | 40 | 40 | 40
Completed | 39 | 38 | 37 | 40 | 39 | 38
Not Completed | 0 | 1 | 2 | 0 | 1 | 2
Not completed — Adverse Event | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of mirikizumab.
Groups:
- Mirikizumab PFS - Abdomen: Participants received 3 mL mirikizumab as 2 SC injections of 1 mL and 2 mL delivered via PFS in the abdomen.
- Mirikizumab AI - Abdomen: Participants received 3 mL mirikizumab as 2 SC injections of 1 mL and 2 mL delivered via AI to the abdomen.
- Total: Total of all reporting groups
Arm/Group | Mirikizumab PFS - Abdomen | Mirikizumab PFS - Arm | Mirikizumab PFS - Thigh | Mirikizumab AI - Abdomen | Mirikizumab AI - Arm | Mirikizumab AI - Thigh | Total
Number analyzed (Participants) | 39 | 39 | 39 | 40 | 40 | 40 | 237
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (12.7) | 39.2 (11.6) | 42.5 (13.2) | 42.1 (14.4) | 42.6 (13.0) | 39.1 (12.8) | 41.3 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 25 | 22 | 21 | 29 | 22 | 138
  Male | 20 | 14 | 17 | 19 | 11 | 18 | 99
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 13 | 8 | 9 | 8 | 48
  Not Hispanic or Latino | 33 | 35 | 26 | 32 | 31 | 32 | 189
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 0 | 0 | 3 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 5 | 5 | 4 | 8 | 3 | 29
  White | 32 | 33 | 33 | 35 | 29 | 36 | 198
  More than one race | 1 | 0 | 1 | 1 | 0 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39 | 39 | 39 | 40 | 40 | 40 | 237

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Mirikizumab Administered by PFS and AI
Description: PK: Cmax of Mirikizumab administered by PFS and AI.
Time Frame: Pre-dose, 72, 120, 192, 264, 360, 528, 696, 1032, 1368, 1704, 2040 hours post day 1 dose
Population: All participants who received at least one dose of mirikizumab and had evaluable PK data. Per protocol, PK analysis were performed to compare all PFS participants together versus all AI participants together.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (μg/mL)
Groups:
- Mirikizumab PFS: Participants received 3 mL mirikizumab as 2 SC injections of 1 mL and 2 mL delivered via PFS to abdomen or arms or thighs.
- Mirikizumab AI: Participants received 3 mL mirikizumab as 2 SC injections of 1 mL and 2 mL delivered via AI to abdomen or arms or thighs.
Arm/Group | Mirikizumab PFS | Mirikizumab AI
Number analyzed (Participants) | 114 | 119
micrograms per milliliter (μg/mL) | 20.0 (44) | 23.5 (40)

2. Primary Outcome: PK: Area Under the Plasma Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞]) of Mirikizumab Administered by PFS and AI
Description: PK: AUC[0-∞] of Mirikizumab administered by PFS and AI.
Time Frame: Pre-dose, 72, 120, 192, 264, 360, 528, 696, 1032, 1368, 1704, 2040 hours post day 1 dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*day per milliliter (μg*day/mL)
Arm/Group | Mirikizumab PFS | Mirikizumab AI
Number analyzed (Participants) | 116 | 120
microgram*day per milliliter (μg*day/mL) | 359 (44) | 412 (39)

3. Primary Outcome: PK: Area Under the Plasma Concentration Versus Time Curve From Time Zero to the Last Measured Concentration Value (AUC[0-tlast]) of Mirikizumab Administered by PFS and AI
Description: PK: AUC[0-tlast] of Mirikizumab administered by PFS and AI.
Time Frame: Pre-dose, 72, 120, 192, 264, 360, 528, 696, 1032, 1368, 1704, 2040 hours post day 1 dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*day per milliliter (μg*day/mL)
Arm/Group | Mirikizumab PFS | Mirikizumab AI
Number analyzed (Participants) | 111 | 117
microgram*day per milliliter (μg*day/mL) | 355 (44) | 411 (38)

ADVERSE EVENTS:
Time Frame: Baseline up to 88 days.
Description: All participants who received at least one dose of mirikizumab. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Arm/Group | Mirikizumab PFS - Abdomen | Mirikizumab PFS - Arm | Mirikizumab PFS - Thigh | Mirikizumab AI - Abdomen | Mirikizumab AI - Arm | Mirikizumab AI - Thigh
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/39 | 0/39 | 0/40 | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/39 | 0/39 | 1/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 8/39 | 13/39 | 8/39 | 13/40 | 9/40 | 9/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Mirikizumab PFS - Abdomen (N=39) | Mirikizumab PFS - Arm (N=39) | Mirikizumab PFS - Thigh (N=39) | Mirikizumab AI - Abdomen (N=40) | Mirikizumab AI - Arm (N=40) | Mirikizumab AI - Thigh (N=40)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0/19 (0) | 0/25 (0) | 0/22 (0) | 1/21 (1) | 0/29 (0) | 0/22 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mirikizumab PFS - Abdomen (N=39) | Mirikizumab PFS - Arm (N=39) | Mirikizumab PFS - Thigh (N=39) | Mirikizumab AI - Abdomen (N=40) | Mirikizumab AI - Arm (N=40) | Mirikizumab AI - Thigh (N=40)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 1 (1) | 6 (11) | 5 (8) | 1 (1)
Pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 3 (3) | 3 (3) | 4 (4) | 4 (4) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 6 (7) | 2 (2) | 1 (1) | 3 (5) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-08-11): https://cdn.clinicaltrials.gov/large-docs/96/NCT05069896/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-28): https://cdn.clinicaltrials.gov/large-docs/96/NCT05069896/SAP_001.pdf